CLINICAL TRIAL: NCT00732173
Title: Survivors of Uterine Cancer Empowered By Exercise and Healthy Diet (SUCCEED)
Brief Title: Exercise and Healthy Diet or Standard Care in Patients in Remission From Stage I or Stage II Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CASE8808; P30CA043703 (NIH); CASE8808 (Other: Case Comprehensive Cancer Center); CASE-8808-CC516 (Other: Cancer Center IRB)
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Counseling; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive a lifestyle intervention, "Survivors of Uterine Cancer Empowered by Exercise and Healthy Diet (SUCCEED)", on a group and individual basis consisting of nutrition, exercise, and behavioral modification counseling from a physician, psychologist, registered dietitian, and physical therapist. Sixteen group sessions will be conducted (10 weekly, 6 bi-weekly) for 6 months. Weight and body mass index, satisfaction with study treatment, and exercise/activity logs are assessed weekly and biweekly. Patients receive additional feedback and support during the weeks not met in a group, including newsletters and telephone and e-mail contact.
  Interventions: Behavioral: behavioral dietary intervention; Behavioral: exercise intervention; Other: counseling intervention; Other: educational intervention; Other: survey administration
- Arm II (Active Comparator): Patients receive usual care informational brochures but no lifestyle counseling related to weight loss, physical activity, and nutrition.
  Interventions: Other: educational intervention

INTERVENTIONS:
Behavioral: behavioral dietary intervention — Undergo SUCCEED lifestyle intervention
  Arms: Arm I
Behavioral: exercise intervention — Undergo SUCCEED lifestyle intervention
  Arms: Arm I
Other: counseling intervention — Undergo SUCCEED lifestyle intervention
  Arms: Arm I
Other: educational intervention — Receive information
Other: survey administration — Undergo SUCCEED lifestyle intervention
  Arms: Arm I

SUMMARY:
RATIONALE: Participating in a diet and exercise program may improve the quality of life of overweight and obese patients who are in remission from endometrial cancer.

PURPOSE: This randomized phase I trial is studying an exercise and healthy diet program to see how well it works compared with standard care in patients in remission from stage I or stage II endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* To reduce morbidity and early mortality in endometrial cancer (EC) survivors through obesity management.

SECONDARY OBJECTIVES:

* To expand and refine a previous pilot study of a behavioral, lifestyle-change education intervention for use in overweight and obese patients in remission from endometrial carcinoma.
* To determine the potential effects and variation of each regimen in these patients.
* To explore potential mediators (self-efficacy, depression) and moderators (body mass index) of healthful dietary and exercise behaviors.
* To evaluate neuronal response to high-versus-low calorie visual food stimuli under fasted (hunger) and fed (satiated) states in brain regions of interest (hypothalamus, lateral orbitofrontal cortex, ventral striatum, insula) using blood oxygenation level dependent (BOLD) functional magnetic resonance imaging (fMRI) before and after a lifestyle (diet and exercise counseling) intervention or usual care in obese EC patients. We will also compare the neuronal responses in obese EC patients to those from normal weight subjects without cancer being seen at the same gynecologic clinic; and, explore modification of the neuronal signals by candidate genes and serum biomarkers in the hypothalamic pituitary-adrenal axis, serotonergic and inflammatory pathways.

OUTLINE: Patients are stratified according to body mass index (25.0-39.9 vs ≥ 40) and randomized to 1 of 2 intervention arms.

* Arm I: Patients receive a lifestyle intervention, "Survivors of Uterine Cancer Empowered by Exercise and Healthy Diet (SUCCEED)", on a group and individual basis consisting of nutrition, exercise, and behavioral modification counseling from a physician, psychologist, registered dietitian, and physical therapist. Sixteen group sessions will be conducted (10 weekly, 6 bi-weekly) for 6 months. Weight and body mass index, satisfaction with study treatment, and exercise/activity logs are assessed weekly and biweekly. Patients receive additional feedback and support during the weeks not met in a group, including newsletters and telephone and e-mail contact.
* Arm II (control): Patients receive usual care informational brochures, but no lifestyle counseling, related to weight loss, physical activity, and nutrition.

Patients undergo physician counseling sessions at baseline and 3, 6, and 12 months. Patients are assessed by weight, anthropometric measures, and body mass index; biomarkers; body composition by dual-energy x-ray absorptiometry/densitometry (DEXA); co-morbidities by the Charlson co-morbidity score; depression by the Beck Depression Inventory (BDI); eating patterns by the Three-Factor Eating Inventory (EI); exercise/physical activity by Leisure Score Index (LSI) and pedometer step count; nutrient intake by 24-hour recall; quality of life by the Functional Assessment of Cancer Therapy-General (FACT-G) and Short-form Medical Outcomes (SF-36); and self-efficacy by the Self-Efficacy Questionnaire (SEQ) and the Weight Efficacy Life-Style (WEL).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I or II (early) endometrial carcinoma

  * Diagnosed within the past 3 years
* Underwent prior surgery consisting of a total abdominal hysterectomy and bilateral salpingo-oophorectomy

  * No evidence of disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* BMI ≥ 25 (overweight/obese)
* Medical clearance from primary care physician
* Approved for contact by treating gynecologic oncologist
* At least a 6th-grade reading level to complete significant reading and homework
* No severe psychiatric illness (e.g., schizophrenia, bipolar disorder) or major depression (Beck Depression Inventory > 29) that needs more aggressive, problem-focused interventions
* No dementia or cognitive deficits
* No pre-existing medical conditions that would be a barrier for participation in unsupervised walking
* No participation in a structured weight loss or exercise program in the past 6 months
* Must agree to and be available for longitudinal follow-up assessments
* Non-English speakers may bring an English-speaking person to all group sessions and visits

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Weight change | at baseline and 3, 6, and 12 months.
  Analysis will be carried out by fitting a mixed model. Weight change will be expressed in terms of absolute and relative weight change. In addition, percent weight change will be calculated. To test the null hypotheses that the groups do not differ in terms of change in weight at 6 or 12 months, parameter estimates from the model will be used to construct subsequent t-test that the difference in means at 3, 6, or 12 months is zero.

SECONDARY OUTCOMES:
Quantitative and qualitative nutrient intake | at baseline and 3, 6, and 12 months.
  24 hour dietary recalls will be conducted using the United States Department of Agriculture (USDA) 5 Step Multiple Pass Method. Information about dietary supplement use will also be obtained. Food intake will be entered into Nutritionist Pro. Fruit/vegetable intake will be assessed using the National Cancer Institute (NCI) All-Day Fruit and Vegetable Screener, which has 10 questions which assess intake of fruits and vegetables during the previous month. A mixed modeling approach will be used.
Minutes spent in moderate and vigorous physical activity | at baseline and 3, 6, and 12 months.
  Assessed with the validated Godin Leisure-Time Exercise questionnaire, a four-item query of usual leisure-time exercise habits. Average frequency of milk, moderate, and strenuous exercise during a typical week are assessed. Duration in minutes of activity along with specific questions regarding walking are included. Complete 7-day pedometer step test at baseline and at 6 and 12 months. A mixed modeling approach will be used.
Body composition, using dual energy x-ray absorptiometry/densitometry (DEXA) methodology | at baseline and 3, 6, and 12 months.
  Measured in a random subsample. Lean body mass, body fat composition, and bone mineral density will be measured. Body composition will be analyzed to determine changes along with weight to help track effectiveness of the intervention.
Biomarkers for metabolic syndrome and nutrition | at baseline and 3, 6, and 12 months.
  Serum biomarkers analyzed for changes along with weight to help track effectiveness of the intervention. Risk factors of metabolic syndrome: low density lipoprotein (LDL), high density lipoprotein (HDL), serum triglycerides, and fasting glucose. Plasma carotenoids (alpha-carotene, beta-carotene, lutein, zeaxanthin) and lycopene concentrations for changes in fruit and vegetable intake. Sub-Study, serum for appetite-related hormones and inflammatory cytokines: leptin, insulin, adiponectin, resistin, IGF-1, IGFBP-1, IGFBP-3, IL-6, TNF-α, MCP-1, glucagon, GLP-1 active, and thyroid hormones.
Self-efficacy | at baseline and 3, 6, and 12 months.
  Self-Efficacy Questionnaire: Physical Activities, an 8 item measure of respondents' perception of the degree to which they feel able to make changes in their physical activity level. Weight Efficacy Life-Style (WEL) questionnaire, 20 questions in 5 situational factors, where subjects rate their ability to successfully resist the desire to eat using a 10-point scale. Methodology of Baron and Kenny used to test for mediating effect of self-efficacy. Multiple regression analyses used to provide statistical tests of the possible mediating role of self-efficacy.
Depression | at baseline and 3, 6, and 12 months.
  Assessed using the Beck Depression Inventory (BDI), a 21-item, Likert-scaled instrument of depressive symptoms. Methodology of Baron and Kenny used to test for mediating effect of depression. Multiple regression analyses used to provide statistical tests of the possible mediating role of depression.
Quality of life | at baseline and 3, 6, and 12 months.
  Using Functional Assessment of Cancer Therapy-General (FACT-G), a 27-item core questionnaire evaluating various domains of QOL including physical, functional, family-social, and emotional well-being with questions answered on a 5-point Likert scale and items summated to give scores for each domain; a 13-item fatigue subscale; and the FACT-Endometrial (En), a 16-item subscale specific for EC. Also using Short-Form (SF)-36, with 36 questions scored on a Likert scale, producing overall physical and mental component summary measures. Baseline scores entered in the regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. Rose, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center; Vivian von Gruenigen, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] von Gruenigen VE, Waggoner SE, Frasure HE, Kavanagh MB, Janata JW, Rose PG, Courneya KS, Lerner E. Lifestyle challenges in endometrial cancer survivorship. Obstet Gynecol. 2011 Jan;117(1):93-100. doi: 10.1097/AOG.0b013e31820205b3. PMID 21173649